CLINICAL TRIAL: NCT01396083
Title: A 6-month Multicenter, Randomized, Double-masked Phase IIIb-study Comparing the Efficacy and Safety of Ranibizumab Intravitreal Injections Versus Dexamethasone Intravitreal Implant in Patients With Visual Impairment Due to Macular Edema Following Central Retinal Vein Occlusion (CRVO)
Brief Title: Efficacy and Safety of Ranibizumab Intravitreal Injections Versus Dexamethasone Intravitreal Implant in Patients With Central Retinal Vein Occlusion (CRVO)
Acronym: COMRADE-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002EDE18; 2011-001020-38 (EudraCT Number)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Visual Impairment; Macular Edema; Central Retinal Vein Occlusion
Keywords: Visual impairment; macular edema; Central retinal vein occlusion; Dexamethasone implant; Ranibizumab
MeSH Terms: conditions — Vision Disorders; Macular Edema; Retinal Vein Occlusion | interventions — Ranibizumab; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab
- Standard of Care (Active Comparator)
  Interventions: Drug: Dexamethasone implant and sham injections

INTERVENTIONS:
Drug: Ranibizumab
  Arms: Ranibizumab
Drug: Dexamethasone implant and sham injections
  Arms: Standard of Care

SUMMARY:
This clinical trial is designed to compare ranibizumab in comparison with Dexamethasone implant® after 6 months of treatment. In the study arm Lucentis will be given monthly in a pro re nata scheme whereas the comparator Dexamethasone implant is given once at Month 0 with sham injections PRN afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with visual impairment due to macular edema following CRVO
* Diagnosis of CRVO at maximum 6 months prior to Screening
* BCVA using ETDRS charts of 20/40 to 20/400 in the study eye

Exclusion Criteria:

* Media clarity, pupillary dilation and patient cooperation not sufficient for adequate fundus photographs
* Central retinal thickness (CRT) < 250 µm in the study eye
* Prior episode of RVO in the study eye
* Active formation of new vessels in the study eye
* Anti-VEGF-treatment in the study or the fellow eye 3 months prior to Baseline
* IOP ≥ 30mmHg or uncontrolled glaucoma; patients may be re-screened after 1 month if they have undergone glaucoma treatment
* Improvement of > 10 letters on BCVA between Screening and Baseline

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (57):
- Germany (36):
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Regensburg, Germany
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Rothenfelde
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg I. Br
  - Novartis Investigative Site, Glauchau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Ingolstadt
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Lauterbach
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Sulzbach
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Würzburg
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Poland (2):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Bytom
- United Kingdom (17):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, Derby
  - Novartis Investigative Site, Gloucester
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Rugby
  - Novartis Investigative Site, Westcliff-on-Sea
  - Novartis Investigative Site, York

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab: Injections consisted of 0.5 mg/0.05 ml solution to be injected intravitreally
- Dexamethasone: Intravitreal implant as per commercial label (700 μg Dexamethasone; long acting release (LAR) over 6 months
Period: Overall Study
Arm/Group | Ranibizumab | Dexamethasone
Started | 124 | 119
Completed | 113 | 72
Not Completed | 11 | 47
Not completed — Adverse Event | 2 | 28
Not completed — Unsatisfactory therapeutic effect | 2 | 13
Not completed — Consent withdrawn | 4 | 5
Not completed — Protocol deviation(s) | 0 | 1
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Administrative problems | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Dexamethasone | Total
Number analyzed (Participants) | 124 | 119 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (11.4) | 66.9 (12.4) | 66.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 46 | 98
  Male | 72 | 73 | 145

OUTCOME MEASURES:

1. Primary Outcome: Mean Average BCVA Change From Month 1 Through Month 6 to Baseline
Description: the average of the changes in BCVA (letters) from baseline to any post-baseline visit, i.e. the mean of six differences to baseline for the six post-baseline visits at month 1 to 6. BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is pproximately 20/20. An increased score indicates improvement in acuity
Time Frame: Baseline, month 6
Population: The Full Analysis Set (FAS) consisted of all patients from the Randomized Set (RS) who had received at least one application of study treatment and had at least one post-baseline assessment for BCVA. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 124 | 119
Letters | 14.6 (11.8) | 4.8 (16.2)

2. Secondary Outcome: Mean BCVA Change at Month 6
Description: The analysis was performed by an analysis of covariance (ANCOVA) model with average change in BCVA (letters) from Visit 1 through Visit 6 as dependent variable, and with the factors center, treatment and covariate baseline BCVA as predictors
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Letters
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 124 | 119
Letters | 14.78 [11.24 to 18.32] | -3.17 [-6.80 to 0.46]

3. Secondary Outcome: Number of Patients Gaining / Losing ≥ 15 / 10 / 5 Letters
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increased score indicates improvement in acuity. This outcome assessed the number of participants who gained 15, 10 or 5 more letters of visual acuity at month 6 as compared with baseline
Time Frame: Baseline, 6 month
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 124 | 119
Participants
  Gain≥15 letters | 73 | 22
  Loss of ≥15 letters | 1 | 31
  Gain ≥10 letters | 89 | 38
  Loss of ≥10 letters | 4 | 35
  Gain ≥5 letters | 104 | 54
  Loss of ≥5 letters | 5 | 40

4. Secondary Outcome: Time to Achieve a Significant Improvement ≥ 15 Letters
Description: The time was analyzed by the Kaplan-Maier-Method, adjusting the calculation for dropouts
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Time to event (Days)
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 124 | 119
Time to event (Days) | 62 [56 to 91] | 98 [63 to NA] — NA - insufficient number of participants with events

5. Secondary Outcome: Change Over Time in BCVA
Description: as for outcome 2
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: letters
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 124 | 119
letters
  Month 1 | 9.77 [7.27 to 12.27] | 9.54 [6.98 to 12.10]
  Month 2 | 12.25 [9.59 to 14.91] | 11.04 [8.31 to 13.76]
  Month 3 | 14.04 [10.92 to 17.16] | 4.99 [1.79 to 8.18]
  Month 4 | 12.76 [9.48 to 16.04] | -1.73 [-5.09 to 1.63]
  Month 5 | 13.57 [10.25 to 16.89] | -2.92 [-6.33 to 0.48]
  Month 6 | 14.78 [11.24 to 18.32] | -3.17 [-6.80 to 0.46]

6. Secondary Outcome: Change Over Time of the Central Retinal Thickness (CRT)
Description: Retinal thickness was measured using Optical Coherence Tomography (OCT). The images were reviewed by a central reading center to ensure a standardized evaluation
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 122 | 119
µm | -376.7 (274.9) | -168.7 (288.3)

7. Secondary Outcome: Changes in the Quality of Life According to the National Eye Institute Visual Function Questionnaire (NEI-VFQ 25) Questionnaires
Description: The VFQ-25 composite and subscale scores range from 0 to 100, a higher score indicating better functioning. The 12 subscales in the VFQ-25 are general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. The scores on the subscales were added together for a total score, which ranged from 0 to 100. A higher score indicated improvement in quality of life due to vision function
Time Frame: Baseline, month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 121 | 118
Score on a scale | 6.0 (12.1) | 2.0 (10.9)

8. Secondary Outcome: Changes in the Quality of Life According to the Short Form (36) Health Survey (SF-36)Questionnaires
Description: SF-36 summary measures are norm-based scores with mean = 50 and SD = 10. Higher scores indicate better health
Time Frame: Baseline, month 6
Population: The Full Analysis Set (FAS) consisted of all patients from the Randomized Set (RS) who had received at least one application of study treatment and had at least one post-baseline assessment for BCVA. observed is only described in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 116 | 113
Units on a scale
  SF-36 physical component (n=116,113) | -0.7 (6.3) | 0.4 (6.6)
  SF-36 mental component (n=116,113) | 2.4 (8.7) | 0.4 (9.2)

9. Secondary Outcome: Changes in the Quality of Life According to Euro Quality of Life (EQ-5D) Questionnaires
Description: The EQ-5D visual analog scale ranges from 0 to 100, 0 representing the worst and 100 the best imaginable health state.
Time Frame: Baseline, month 6
Population: The Full Analysis Set (FAS) consisted of all patients from the Randomized Set (RS) who had received at least one application of study treatment and had at least one post-baseline assessment for BCVA. Observed participants are only described in this analysis
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 116 | 113
Units on a scale | 0.1 (13.2) | 2.0 (14.8)

10. Secondary Outcome: Increase Rate of the Internal Ocular Pressure (IOP ) : Patients With ≥10% Increase in IOP Compared to Baseline
Description: The proportion of patients with ≥ 10% increase in Internal Ocular Pressure (IOP) compared to baseline at any post-baseline visit.
Time Frame: Baseline, month 6
Population: The Safety Set consisted of all patients from the RS who had received at least one application of study treatment and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received. The statement that a patient had no adverse events also constituted a safety assessment
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Dexamethasone
Number analyzed (Participants) | 124 | 119
Participants | 94 | 105

ADVERSE EVENTS:
Arm/Group | Ranibizumab | Dexamethasone
Serious Adverse Events (participants affected / at risk) | 10/124 | 16/119
Other Adverse Events (participants affected / at risk) | 77/124 | 99/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=124) | Dexamethasone (N=119)
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1
ADENOMATOUS POLYPOSIS COLI (Congenital, familial and genetic disorders) | 1 | 0
DEAFNESS (Ear and labyrinth disorders) | 0 | 1
CONJUNCTIVAL HYPERAEMIA (Study eye) (Eye disorders) | 0 | 1
CORNEAL OEDEMA (Study eye) (Eye disorders) | 0 | 1
EYE PAIN (Study eye) (Eye disorders) | 0 | 1
GLAUCOMA (Study eye) (Eye disorders) | 0 | 3
HYPHAEMA (Study eye) (Eye disorders) | 0 | 3
IRIS NEOVASCULARISATION (Study eye) (Eye disorders) | 0 | 4
MACULAR OEDEMA (Study eye) (Eye disorders) | 1 | 2
RETINAL ARTERY OCCLUSION (Study eye) (Eye disorders) | 0 | 1
RETINAL VEIN OCCLUSION (Study eye) (Eye disorders) | 1 | 1
VISUAL ACUITY REDUCED (Study eye) (Eye disorders) | 0 | 3
VITREOUS HAEMORRHAGE (Study eye) (Eye disorders) | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1
GASTRODUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
CYSTITIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INTRAOCULAR PRESSURE DECREASED (Study eye) (Investigations) | 0 | 1
INTRAOCULAR PRESSURE INCREASED (Study eye) (Investigations) | 0 | 1
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1
RADIAL NERVE PALSY (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 2
PROSTATITIS (Reproductive system and breast disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=124) | Dexamethasone (N=119)
ABNORMAL SENSATION IN EYE (Study eye) (Eye disorders) | 6 | 8
CONJUNCTIVAL HAEMORRHAGE (Study eye) (Eye disorders) | 16 | 13
DRY EYE (Fellow eye) (Eye disorders) | 4 | 1
DRY EYE (Study eye) (Eye disorders) | 4 | 4
EYE IRRITATION (Study eye) (Eye disorders) | 4 | 3
EYE PAIN (Study eye) (Eye disorders) | 15 | 14
FOREIGN BODY SENSATION IN EYES (Study eye) (Eye disorders) | 6 | 6
GLAUCOMA (Study eye) (Eye disorders) | 0 | 5
IRIS NEOVASCULARISATION (Study eye) (Eye disorders) | 0 | 5
LACRIMATION INCREASED (Study eye) (Eye disorders) | 6 | 8
MACULAR ISCHAEMIA (Study eye) (Eye disorders) | 0 | 3
MACULAR OEDEMA (Study eye) (Eye disorders) | 13 | 19
OCULAR HYPERAEMIA (Study eye) (Eye disorders) | 14 | 15
OCULAR HYPERTENSION (Study eye) (Eye disorders) | 0 | 6
OPTIC DISC VASCULAR DISORDER (Study eye) (Eye disorders) | 5 | 0
RETINAL EXUDATES (Study eye) (Eye disorders) | 2 | 4
RETINAL ISCHAEMIA (Study eye) (Eye disorders) | 1 | 6
RETINAL VASCULAR DISORDER (Study eye) (Eye disorders) | 2 | 5
VISUAL ACUITY REDUCED (Study eye) (Eye disorders) | 8 | 19
VISUAL IMPAIRMENT (Study eye) (Eye disorders) | 2 | 6
VITREOUS DETACHMENT (Study eye) (Eye disorders) | 5 | 3
VITREOUS FLOATERS (Study eye) (Eye disorders) | 5 | 11
DIARRHOEA (Gastrointestinal disorders) | 6 | 2
NAUSEA (Gastrointestinal disorders) | 4 | 3
PYREXIA (General disorders) | 0 | 3
BRONCHITIS (Infections and infestations) | 1 | 3
NASOPHARYNGITIS (Infections and infestations) | 9 | 12
URINARY TRACT INFECTION (Infections and infestations) | 1 | 4
BLOOD GLUCOSE INCREASED (Investigations) | 4 | 2
INTRAOCULAR PRESSURE INCREASED (Fellow eye) (Investigations) | 0 | 3
INTRAOCULAR PRESSURE INCREASED (Study eye) (Investigations) | 7 | 38
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 4
HEADACHE (Nervous system disorders) | 7 | 10
HYPERTENSION (Vascular disorders) | 5 | 3
VASCULAR SHUNT (Study eye) (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety